CLINICAL TRIAL: NCT03004365
Title: A Phase 2, Single-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Microbiology of C16G2 Varnish Administered in Multiple Doses to Adolescent and Adult Dental Subjects
Brief Title: A Study to Evaluate the Safety and Microbiology of C16G2 Varnish Administered in Multiple Doses to Dental Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: C3J16-V204-00
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1A: 27.2 mg C16G2 (Active Comparator): Subjects in Study Arm 1 will receive up to 1 mL of 27.2 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: C16G2 Varnish
- Arm 1B: 27.2 mg Placebo (Placebo Comparator): Subjects in Study Arm 1 will receive up to 1 mL of 27.2 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: Placebo Varnish
- Arm 2A: 13.6 mg C16G2 (Active Comparator): Subjects in Study Arm 2 will receive up to 1 mL of 13.6 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: C16G2 Varnish
- Arm 2B: 13.6 mg Placebo (Placebo Comparator): Subjects in Study Arm 2 will receive up to 1 mL of 13.6 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: Placebo Varnish
- Arm 3A: 54.4 mg C16G2 (Active Comparator): Subjects in Study Arm 3 will receive up to 1 mL of 54.4 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: C16G2 Varnish
- Arm 3B: 54.4 mg Placebo (Placebo Comparator): Subjects in Study Arm 3 will receive up to 1 mL of 54.4 mg C16G2 Varnish or Placebo Varnish on day 1, followed by two additional applications a week and two weeks later, for a total of 3 study drug applications. Study drug will be administered via a small brush typically used in varnish applications.
  Interventions: Drug: Placebo Varnish

INTERVENTIONS:
Drug: C16G2 Varnish — Antimicrobial Peptide
  Arms: Arm 1A: 27.2 mg C16G2; Arm 2A: 13.6 mg C16G2; Arm 3A: 54.4 mg C16G2
Drug: Placebo Varnish — Placebo
  Arms: Arm 1B: 27.2 mg Placebo; Arm 2B: 13.6 mg Placebo; Arm 3B: 54.4 mg Placebo

SUMMARY:
The purpose of this single-blind study is to evaluate whether C16G2 Varnish administered in multiple doses can effectively kill the bacteria in the oral cavity that cause dental caries.

DETAILED DESCRIPTION:
A single-blind, randomized, placebo-controlled Phase 2 study to evaluate the safety and oral microbiology of C16G2 Varnish application in male and female dental subjects 12-75 years of age. This multi-center study will evaluate multiple study drug administrations of C16G2 Varnish or Placebo Varnish.

The study will enroll subjects into up to three study arms. Up to 33 subjects will receive multiple doses of study drug applied with a small brush typically used in dental varnish administration. Subjects will be enrolled in an 8:3 ratio. The Sponsor will perform unblinded microbiology review on an ongoing basis to determine whether to enroll additional 11 subjects into the next dose cohort or to terminate enrollment based on microbiology data.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 12-75 years of age
2. Adults subjects provide written informed consent and adolescent subjects give written or verbal assent, as appropriate, and parent(s) or legal guardian(s) give written informed consent
3. Female subjects of childbearing potential must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, relationship with a same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
4. Negative urine pregnancy test in all females of childbearing potential (past menarche)
5. Male subjects of sexual activity age: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
6. Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (general, extraoral, head and neck) during Screening.

   Note: Subjects on a stable dose of medication may be eligible for screening and will be assessed by the medical monitor on a case-by-case basis.
7. Have a minimum of 12 bicuspids and molars with a minimum of 8 molars and bicuspids NOT having restorations, crowns or sealants
8. Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
9. Have a salivary S. mutans of 1.0 x 10^5 CFUs/mL or greater at Screening using mitis salivarius-bacitracin (MSB) agar plating
10. Willing to refrain from using non-study dentifrice and other non-study oral care products (oral care rinses, fluoride products, etc.) during the study
11. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
12. Willing and able to comply with oral hygiene and diet instructions
13. Able to communicate with the Investigator/study center personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by comprehensive caries examination including standard radiographs). Subjects presenting with insipient, non-cavitated lesion(s) are not excluded.

   Note: If radiographs are deemed appropriate for the study and taken within 6 months prior to the Screening visit, these may be used for determining eligibility and not required to be repeated at Screening
3. Partially erupted teeth where the entire crown is not erupted or an operculum is present
4. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
5. Pathologic lesions of the oral cavity (suspicious or confirmed)
6. Full dentures or permanent orthodontic appliances, e.g., braces, buccal or lingual brackets. Note: Partial dentures, removable retainers and night guards are not excluded, provided that they are cleaned regularly throughout the duration of the study
7. Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, beginning 30 days prior to Screening until the end of study participation
8. Medical history indicating the woman is pregnant, breastfeeding/lactating or has a positive urine pregnancy test
9. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
10. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pittaway, DMD, Principal Investigator — Plaza West II Dental Group
Locations (3):
- United States (3):
  - John F. Pittaway, DMD, Kalispell, Montana
  - Jacqueline Kleven, DDS, Bedford, Texas
  - Anthony Henegar, DDS, PA, Irving, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Group: Pooled Placebo: Subjects enrolled in Arms 1B (N=3), 2B (N=3) and 3B (N=3) were pooled into one group.
Period: Overall Study
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo
Started | 8 | 8 | 8 | 9
Completed | 8 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 33
Age, Continuous [Mean (Full Range); unit: years] | 28.7 [18 to 53] | 28.7 [14 to 52] | 19.4 [17 to 24] | 22.2 [16 to 54] | 24.7 [14 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 6 | 21
  Male | 2 | 3 | 4 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 4 | 4 | 10
  Not Hispanic or Latino | 6 | 8 | 4 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Safety of Multiple C16G2 Varnish Applications
Description: Safety will be assessed by performing targeted physical examinations, oral cavity exams, taking vital signs and collection of adverse events categorized according to system organ class (SOC) and preferred term (PT) based on coding to the Medical Dictionary for Regulatory Activities (MedDRA®), Version 17.1. Comprehensive examinations of oral hard and soft tissue structures, as well as targeted exams of specific musculoskeletal and extraoral sites were performed at selected time points; vital signs (blood pressure, heart rate and temperature) were taken at screening, baseline (Visit 3/Day 0) and Visits 4 and 5.
Time Frame: Subjects will be followed for safety for 1 week post last study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
Participants
  Participants with Adverse Events Related to Study Drug | 0 | 0 | 0 | 0
  Participants with Clinical Significant Oral Cavity Changes | 0 | 0 | 0 | 0
  Participants with Clinical Significant Vital Sign Changes | 0 | 0 | 0 | 0
  Participants with Abnormal Physical Exam Findings | 0 | 0 | 0 | 0
  Participants with Completed Study | 8 | 8 | 8 | 9

2. Secondary Outcome: Antimicrobial Activity Against S. Mutans
Description: To assess the targeted antimicrobial activity of C16G2 applications as measured by a reduction in Streptococcus mutans in saliva and dental plaque using S. mutans CFUs using mitis-salivarius bacitrain (MSB) agar plating. Streptococcus species present in the oral cavity have been traditionally isolated from oral cavity samples using MSB agar plates. A summary focusing on mean log transformed S. mutans changes from baseline levels in saliva at each assessment time point following the first administration of C16G2.The log transformed changes from baseline S. mutans levels in saliva at each assessment time point following the first administration of C16G2 in each study arm including N, mean, SD, median and range.
Time Frame: Subjects will be followed for microbiology for 1 month post last study drug administration
Measure: Mean (Standard Deviation); unit: log(CFU/mL)
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
log(CFU/mL)
  Saliva Sample: S. mutans by MSB Agar Plating | -0.23 (0.60) | -0.08 (0.54) | -0.015 (0.63) | -0.09 (0.46)
  Dental Plaque: S. mutans by MSB Agar Plating | -0.51 (0.8) | -0.28 (0.54) | -0.58 (0.6) | -0.59 (0.74)

3. Secondary Outcome: Antimicrobial Activity Against Total Bacteria
Description: To assess total bacteria in saliva and dental plaque post study drug administration using total bacteria CFUs using Todd Hewitt (TH) agar plating and the log transformed changes from baseline Total Bacteria levels in dental plaque and saliva including N, mean, SD, median and range at each assessment time point following the first administration of C16G2. A summary focusing on mean log transformed S. mutans changes from baseline levels in saliva at each assessment time point following the first administration of C16G2.
Time Frame: Subjects will be followed for microbiology for 1 month post last study drug administration
Measure: Mean (Standard Deviation); unit: log(CFU/mL)
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 9
log(CFU/mL)
  Saliva Sample - Total Bacteria by TH Agar Plating | 0.21 (0.49) | -0.03 (0.22) | -0.09 (0.55) | 0.07 (0.22)
  Dental Plaque - Total Bacteria by TH Agar Plating | -0.46 (0.69) | -0.58 (0.3) | -0.51 (0.57) | -0.24 (0.56)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Arm 1A: 27.2 mg C16G2 | Arm 2A: 13.6 mg C16G2 | Arm 3A: 54.4 mg C16G2 | Group: Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03004365/Prot_SAP_000.pdf